CLINICAL TRIAL: NCT07332754
Title: Retrospective Observational Study on the Use of Advanced Bacterial-binding Dressings (DACC-coated Hydrogel Dressings) in Radiodermatitis in Women Undergoing Radiotherapy for Breast Cancer
Brief Title: Retrospective Observational Study on the Use of Advanced Bacterial-binding Dressings (DACC-coated Hydrogel Dressings) in Radiodermatitis
Acronym: RadioDACC
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: RadioDACC
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Radiodermatitis; Acute
Keywords: radiodermatitis; acute wound care treatment; DACC-coated hydrogel dressing; radiotherapy; breast cancer
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Female patients undergoing adjuvant radiotherapy affected by radiodermatitis for breast cancer: Female patients treated with a DACC-coated hydrogel device following the diagnosis of grade 2-3 radiodermatitis according to the RTOG scale mainly localized in the inframammary region, with or without axillary or supraclavicular extension.
  Outpatient treatment with an advanced dressing protocol including: cleansing with 0.05% sodium hypochlorite solution, application of DACC-coated hydrogel dressing with replacement every 2-3 days.

SUMMARY:
the study aimed to evaluate the clinical effectiveness, safety and tolerability of a DACC-coated hydrogel advanced dressing for the treatment of radiodermatitis in patients undergoing radiotherapy for breast cancer.

DETAILED DESCRIPTION:
The planned assessments include recording RTOG and NRS scores at time points T0 (starting treatment), T1, and T2 (end of treatment), documenting the time to complete re-epithelialization, any interruption of radiotherapy treatment, and collecting organizational and economic data for HTA and SWOT analyses.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age ≥18 years
* Histologically confirmed diagnosis of breast cancer, undergoing adjuvant radiotherapy after surgery and/or chemotherapy.
* Onset of grade 2-3 radiodermatitis according to the RTOG scale, mainly located in the inframammary region, with or without axillary or supraclavicular extension.
* Patients treated with a DACC-coated hydrogel device following a radiodermatitis diagnosis, between January 2023 and October 2025.
* Treated on an outpatient basis with an advanced dressing protocol including:

  * Cleansing with 0.05% sodium hypochlorite solution
  * Application of DACC-coated hydrogel dressing, replaced every 2-3 days.
* Complete clinical data available in outpatient records, including NRS and RTOG.

Exclusion Criteria:

* Grade 0 radiodermatitis (absence of skin toxicity)
* Patients with incomplete clinical data or insufficient documentation for the purposes of retrospective analysis
* Lack of availability of minimum clinical follow-up until complete re-epithelialization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: The study population includes adult female patients (≥18 years) with histologically confirmed breast cancer who underwent adjuvant radiotherapy at IRCCS Ospedale Galeazzi Sant'Ambrogio (Milan, Italy) between January 2023 and October 2025 and developed acute radiation dermatitis requiring treatment. Most patients presented with moderate to severe radiation dermatitis (RTOG grade 2-3), predominantly involving the inframammary region, with or without axillary or supraclavicular extension. A limited number of patients with grade 1 dermatitis were also included when clinically justified, in order to reflect real-world clinical practice. All patients were managed in an outpatient setting using a standardized protocol with a DACC-coated hydrogel dressing, and complete clinical documentation was available for retrospective analysis.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of clinical effectiveness of the advanced DACC-coated hydrogel dressing | From enrollment to the end of treatment at T2 (clinical resolution/complete re-epithelialization within 20 days from the start of treatment (T0).
  Evaluate the clinical effectiveness of the advanced DACC-coated hydrogel dressing used in the management of severe radiodermatitis in patients undergoing radiotherapy for breast cancer; effectiveness will be measured by assessing the reduction in pain using the NRS at the beginning and end of the treatment (from T0 to T2).

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Ospedale Galeazzi Sant'Ambrogio, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No
Not applicable. Individual participant data will not be shared, as this is a retrospective, single-center observational study based on routinely collected clinical data that are pseudonymized and subject to institutional and regulatory privacy restrictions.